CLINICAL TRIAL: NCT04845711
Title: Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Cholecystectomy Surgeries: A Randomized Controlled Trial
Brief Title: Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Elsaid Hamada, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34503/2/21
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Analgesia; Erector Spinae Plane Block; Quadratus Lumborum Block
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and medical personnel collecting data and conducting follow-up will be blinded to the group of the patient. All blocks will be performed by one anesthesiologist who will not participate in data collection or analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): patients will receive general anesthesia only.
  Interventions: Other: Control group
- Erector spinae plane block group (Experimental): patients will receive general anesthesia and bilateral ultrasound guided erector spinae plane block (20ml Bupivacaine 0.25%)
  Interventions: Procedure: Erector spinae plane block group
- Quadratus lumborum block group (Experimental): patients will receive general anesthesia and bilateral ultrasound guided quadratus lumborum block (20 ml Bupivacaine 0.25%)
  Interventions: Procedure: Quadratus lumborum block group

INTERVENTIONS:
Other: Control group — patients will receive general anesthesia only.
  Other Names: Group C
  Arms: Control group
Procedure: Erector spinae plane block group — patients will receive general anesthesia and bilateral ultrasound guided erector spinae plane block (20ml Bupivacaine 0.25%)
  Other Names: group ESPB
  Arms: Erector spinae plane block group
Procedure: Quadratus lumborum block group — patients will receive general anesthesia and bilateral ultrasound guided quadratus lumborum block (20 ml Bupivacaine 0.25%)
  Other Names: group QLB
  Arms: Quadratus lumborum block group

SUMMARY:
The aim of this study is to compare between the efficacy of ultrasound guided erector spinae plane block and ultrasound guided quadratus lumborum block in managing acute postoperative pain in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-65 years
* both genders
* American Society of Anesthesiology (ASA) class I-II
* Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patient refusal.
* Coagulopathy.
* History of allergy to local anaesthetic.
* History of liver or renal pathology affecting drug elimination
* Mental dysfunction or cognitive disorders.
* Use of medication such as gabapentin-pregabalin that could affect pain perception.
* Body Mass Index > 40 kg/m2.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
The degree of postoperative pain in the first 24 hours post-operative | first 24 hours post-operative
  Postoperative pain will be assessed by the numerical rating scale (NRS); 0 no pain while 10 is the maximum pain) after discharge to the ward ,and at 6, 12, 18, 24 hours.

SECONDARY OUTCOMES:
Time to first analgesic requirement | first 24 hours post-operative
  Intravenous morphine 2 mg will be given when the numerical rating scale (NRS) equal or above 4
Total dose of intraoperative consumption of fentanyl | intraoperative
  Fentanyl 0.5 μg/kg will be given if there was increase in heart rate or mean arterial blood pressure more than 20% (after exclusion of other causes than pain).
Total dose of rescue analgesia in the first 24hr postoperative | first 24 hours post-operative
  Total morphine consumption 24 hours after surgery will be recorded. Intravenous morphine 2 mg will be given when the numerical rating scale (NRS) equal or above 4

CONTACTS AND LOCATIONS:
Overall Officials: Mai E Hamada, MBBCH, Principal Investigator — Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after the end of study For 2 years
Access Criteria: Data are available upon reasonable request from the principal investigator